CLINICAL TRIAL: NCT01528124
Title: A Single-Dose, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of LY3025876 in Healthy Subjects
Brief Title: A Study of LY3025876 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14346; I6D-FW-SMRA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% sodium chloride given as a single subcutaneous injection
  Interventions: Drug: Placebo
- LY3025876 (Experimental): Single escalating doses of LY3025876 given as subcutaneous injections
  Interventions: Drug: LY3025876

INTERVENTIONS:
Drug: LY3025876 — Given as a subcutaneous injection
  Arms: LY3025876
Drug: Placebo — Given as a subcutaneous injection
  Arms: Placebo

SUMMARY:
This trial is conducted in Singapore. The aim of this trial is to evaluate the safety and tolerability of the study drug in healthy people and investigate how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Must be either a healthy male or a healthy female who cannot become pregnant
* Have a body mass index (BMI) of 18.5 to 40.0 kilograms per meter squared (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Are allergic to LY3025876 or related compounds
* Have a history of significant disease that may affect the actions of drugs or may pose a risk when taking the study medication
* Have a history of developing allergies, asthma, severe drug allergies (symptoms including, but not limited to, itching, red rashes, sores on the skin, scaling and shedding of skin), allergies or reactions to more than one drug, or have had bad reactions to skin creams containing corticosteroids. Corticosteroids are mainly used to control inflammation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Normal sterile saline solution (0.9% sodium chloride) administered as subcutaneous injection
- 0.15 mg LY3025876: 0.15 milligrams (mg) LY3025876 administered as subcutaneous injection
- 0.5 mg LY3025876: 0.5 mg LY3025876 administered as subcutaneous injection
- 1.5 mg LY3025876: 1.5 mg LY3025876 administered as subcutaneous injection
- 5 mg LY3025876: 5 mg LY3025876 administered as subcutaneous injection
- 15 mg LY3025876: 15 mg LY3025876 administered as subcutaneous injection
- 30 mg LY3025876: 30 mg LY3025876 administered as subcutaneous injection
Period: Overall Study
Arm/Group | Placebo | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Started | 6 | 6 | 6 | 6 | 5 | 6 | 6
Received Study Drug | 6 | 6 | 6 | 6 | 5 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.9) | 36.8 (8.8) | 33.7 (9.3) | 32.7 (3.8) | 29.4 (7.4) | 27.8 (4.5) | 31.3 (7.2) | 32.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Male | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 41
Fasting Blood Glucose [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 4.68 (0.17) | 4.45 (0.40) | 4.43 (0.40) | 4.97 (0.27) | 4.68 (0.33) | 4.20 (0.35) | 4.57 (0.36) | 4.57 (0.38)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per meter squared (kg/m^2)] | 28.35 (2.31) | 23.88 (4.91) | 26.22 (5.65) | 25.12 (1.99) | 26.78 (6.62) | 23.10 (3.48) | 25.53 (2.91) | 25.54 (4.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Drug-related Adverse Events or Any Serious Adverse Events
Description: Possible drug-relatedness of an adverse event (AE) was in the opinion of the investigator. A summary of all serious and all other non-serious AEs, regardless of any possible causality, is located in the Reported Adverse Event Module.
Time Frame: Baseline up to 28 days post-dose
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6 | 6
participants
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other nonserious AEs | 0 | 0 | 1 | 1 | 1 | 0 | 1

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3025876
Description: Area under the concentration-versus-time curve from time zero to infinity [AUC(0-∞)] of LY3025876.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose
Population: Pharmacokinetic (PK) Population: all participants who received at least 1 dose of study drug and had evaluable AUC(0-∞) PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Number analyzed (Participants) | 6 | 5 | 6 | 5 | 6 | 6
nanograms*hour per milliliter (ng*h/mL) | NA (NA) — Not calculated, insufficient LY3025876 plasma concentrations were quantifiable for calculating AUC. | 62.5 (11.9) | 180 (17.0) | 595 (8.74) | 1920 (9.99) | 3780 (25.1)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3025876
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours post-dose
Population: PK Population: all participants who received at least 1 dose of study drug and had evaluable Cmax PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
nanograms per milliliter (ng/mL) | 1.88 (35.2) | 7.25 (53.1) | 16.0 (18.2) | 55.0 (26.5) | 187 (22.9) | 347 (19.6)

4. Secondary Outcome: Number of Participants Developing Anti-LY3025876 Antibodies
Description: Blood samples were collected from all randomized participants to test for the development of antibodies binding to LY3025876.
Time Frame: Day 28 post-dose
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | 0.15 mg LY3025876 | 0.5 mg LY3025876 | 1.5 mg LY3025876 | 5 mg LY3025876 | 15 mg LY3025876 | 30 mg LY3025876
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 2/6 | 3/6 | 1/6 | 2/5 | 3/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | 0.15 mg LY3025876 (N=6) | 0.5 mg LY3025876 (N=6) | 1.5 mg LY3025876 (N=6) | 5 mg LY3025876 (N=5) | 15 mg LY3025876 (N=6) | 30 mg LY3025876 (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Application site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes